CLINICAL TRIAL: NCT05614752
Title: A Multi-Center, Prospective, Observational Study to Evaluate the Improvement Effect on Subjective Symptom of FEXUCLUE Tab. in Patients With Erosive Gastroesophageal Reflux Disease
Brief Title: Study to Evaluate the Improvement Effect on Subjective Symptom of FEXUCLUE Tab
Status: Completed | Type: Observational
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Other Study IDs: DWFE_P406
Record Dates: First submitted 2022-11-07; First posted 2022-11-14 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — fexuprazan

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment group: treated with Fexuclue Tablet 40mg
  Interventions: Drug: Fexuprazan

INTERVENTIONS:
Drug: Fexuprazan — Fexuclue Tablet 40mg

SUMMARY:
This observational study is a large-scale, prospective, and multi-institutional observational study.

Patients from 19 to 75 years of age, will take a self-assessment (PRO) during the study period before and after administration of Pexuclue tablet.

DETAILED DESCRIPTION:
Data will be collected based on patient's medical records from daily visit. Enrolled subjects will take a Patient Reported Outcome (PRO) survey including Quality of life evaluation (GERD-HRQL) and self-awareness symptom (RDQ).

The survey will be done twice (before and after the administration of Fexuclue tablet) electronically through an application (e-PRO).

ELIGIBILITY:
Inclusion Criteria:

1. Adult aged 19 years to 75 years (on registration date)
2. Patient scheduled to administer Fexuclue tablet based on the medical judgment of investigator.
3. Patient who agreed to participate in this observation study and signed Informed Consent Form

Exclusion Criteria:

1. A person who falls under the prohibition of administration according to the permission for Fexuclue Tablet

   * Patients with hypersensitivity to the components of Fexuclue tablet or Fexuclue tablet and a history thereof
   * Patients undergoing Atazanavir, Nelfinavir or Lilpivirin-containing preparations
   * Pregnant and lactating women
   * Patients with genetic problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabortion
2. A person who participates in another clinical trial and is administering (applying) clinical trial drugs or clinical trial medical devices;
3. In addition to the above, a person who has determined that the researcher (the doctor in charge) is not suitable for participation in this observation study

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population was calculated by the average of changes and standard deviation at two weeks and by referring to Michael Shaw et al. (2008)'s RDQ score (reverse flow, heartburn, indigestion)
Sampling Method: Probability Sample
Enrollment: 10067 (Actual)
Dates: Start 2022-07-06 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-11-08 (Actual)

PRIMARY OUTCOMES:
Average score change in RDQ | At least 2 weeks (up to 8 weeks)
  Average score change in RDQ at least 2 weeks (up to 8 weeks) compared to baseline

SECONDARY OUTCOMES:
changes in average score of the individual symptoms (reflux, heartburn, indigestion) | At least 2 weeks (up to 8 weeks)
  changes in average score of the individual symptoms (reflux, heartburn, indigestion) at least 2 weeks(up to 8 weeks) from baseline (0~5)
RDQ validity rate | At least 2 weeks (up to 8 weeks)
  RDQ validity rate at least 2 weeks(up to 8 weeks) from baseline
Overall improvement evaluated by the subjects | At least 2 weeks (up to 8 weeks)
  Overall improvement result (scale 1~5, Fully recovered/Much improvement/Moderate improvement/Unchanged/Aggravated) evaluated by the subjects at least 2 weeks(up to 8 weeks) from baseline
Overall improvement evaluated by the researchers | At least 2 weeks (up to 8 weeks)
  Overall improvement (scale 1~5, Fully recovered/Much improvement/Moderate improvement/Unchanged/Aggravated) evaluated by the researchers at least 2 weeks(up to 8 weeks) from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Seungyoung Seo, Principal Investigator — Jeonbuk National University Hospital
Locations (1):
- Jeonbuk National University Hospital, Jeonju, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
Not yet decided